CLINICAL TRIAL: NCT05456789
Title: A Randomized Trial for Catheter-interventional Treatment of Intermediate High Risk Pulmonary Embolism
Brief Title: Catheter-interventional Treatment of Pulmonary Embolism
Acronym: CATCH-PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CATCH-PE
Record Dates: First submitted 2022-06-16; First posted 2022-07-13 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined interventional treatment (Experimental): Combined catheter-based fibrinolysis and thrombectomy plus conventional treatment
  Interventions: Device: combined catheter-thrombectomy and local fibrinolysis
- conventional treatment (Active Comparator): Conventional treatment
  Interventions: Other: conventional treatment

INTERVENTIONS:
Device: combined catheter-thrombectomy and local fibrinolysis — combination of catheter-based thrombectomy with local pulmonary fibrinolysis plus conventional treatment
  Arms: Combined interventional treatment
Other: conventional treatment — conventional treatment of pulmonary embolism
  Arms: conventional treatment

SUMMARY:
Recent evidence supports the use of catheter-interventional techniques for the treatment of intermediate-high-risk pulmonary embolism. While there is evidence supporting the use of catheter-thrombectomy and alternatively local fibrinolysis, less is known on the combination of both approaches.

The investigators aim to assess the effects of a combined interventional local fibrinolysis and catheter-thrombectomy and to compare them with conventional treatment in a cohort of patients with intermediate-high-risk pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* confirmed intermediate high-risk pulmonary embolism
* age >= 18 years

Exclusion Criteria:

* high-risk pulmonary embolism
* contraindications for catheter-based treatment
* known allergy to anticoagulant treatment or fibrinolytics
* pregnancy
* participation in other randomized trials
* patients under legal supervision or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
RV-LV-Ratio | Day 1 after randomization
  Change in right to left ventricular diameter ratio
clinical efficacy | Day 1 after randomization
  quotient of systolic systemic blood pressure over heart rate and respiratory rate

SECONDARY OUTCOMES:
Mortality | 1 day, 30 days, 1 year after randomization
  difference in mortality between the treatment groups
Right heart failure | 30 days and 1 year after randomization
  difference in new onset right heart failure between the groups
pulmonary artery pressure | 1 day, 30 days and 1 year after randomization
  difference in estimated pulmonary artery pressure between the groups
RV/LV-ratio | 30 days and 1 year after randomization
  difference in RV/LV-ratio
TAPSE | 1 day, 30 days and 1 year after randomization
  difference in TAPSE as assessed by transthoracic echocardiogram
difference in RA volume between the groups | 1 day, 30 days and 1 year after randomization
  RA volume between the groups
Bleeding | 1 day, 30 days and 1 year after randomization
  difference in BARC bleeding events between the groups
Troponin and NT-proBNP | 30 days and 1 year after randomization
  difference in high-sensitivity Troponin T and NT-proBNP between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center Leipzig at University of Leipzig, Leipzig, Saxony, Germany